CLINICAL TRIAL: NCT07122453
Title: A Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Single Ascending Doses of Intrathecal CNTX-3001 in Subjects With Intractable Chronic Moderate to Severe Low Back Pain
Brief Title: Safety and PK of Intrathecal CNTX-3001 for Intractable Chronic Low Back Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNTX-3001it-LBP-101; 1UG3NS123965-01 (NIH)
Record Dates: First submitted 2025-07-03; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CNTX-3001 (Experimental): Single intrathecal injection of CNTX-3001
  Interventions: Drug: CNTX-3001
- Placebo (Placebo Comparator): Single intrathecal injection of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTX-3001 — non-opioid analgesic
  Arms: CNTX-3001
Drug: Placebo — Placebo product
  Arms: Placebo

SUMMARY:
This clinical study is being conducted to evaluate the safety, tolerability, plasma pharmacokinetics and efficacy of an investigational drug called CNTX-3001. This Phase 1 study is the first time that CNTX-3001 will be given to people (first-in-human study). The study is being done to evaluate whether CNTX-3001, given into the intrathecal space by lumbar puncture, can be administered safely to participants who have been diagnosed with intractable chronic moderate to severe low back pain and who have not responded well to other treatments in the past.

CNTX-3001 is a novel, non-opioid small molecule

ELIGIBILITY:
Inclusion:

* Have stable intractable, chronic moderate to severe low back pain
* Must have failed all 3 of the following categories of therapies:

  1. Physical medicine modalities for at least 6 weeks (e.g., physical therapy, occupational therapy, or chiropractic treatment directed at chronic low back pain)
  2. Three or more classes of pharmacologic treatments
  3. One or more non-surgical and/or surgical interventions addressing the primary cause of chronic low back pain
* If the intractable low back pain is accompanied by radicular pain, back pain must be dominant over leg pain and may not radiate below the knee
* Has normal leg strength in both legs (able to stand/walk)
* Willing and able to undergo the lumbar puncture
* On a stable analgesic regimen, or a stable dose of an opioid medication for >3 months
* Non- or ex-smoker and has not used any nicotine-containing products within 3 months
* Men or women able to abide by reproductive and contraceptive requirements
* Has a body mass index (BMI) between 18 and 35 kg/m2, with weight ≥60 kg

Exclusion

* Substantial increase or decrease in pain over the prior 3 months.
* Low back pain that only occurs with specific activities or body positions.
* Has asthma or other severe respiratory disease requiring daily prescription medication
* History of, or current cancer (except basal cell carcinoma), cardiac disease, immunological disorders, meningitis, or bleeding disorders
* Confirmed diagnosis of fibromyalgia or myalgic encephalomyelitis

Exclusion

* Substantial increase or decrease in pain over the prior 3 months
* Low back pain that only occurs with specific activities or body positions
* Has asthma or other severe respiratory disease requiring daily prescription medication
* History of, or current cancer (except basal cell carcinoma), cardiac disease, immunological disorders, meningitis, or bleeding disorders
* Confirmed diagnosis of fibromyalgia or myalgic encephalomyelitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | From baseline to the end of treatment visit (Day 7)
  Number of participants with TEAEs, which includes laboratory test variables

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of CNTX-3001 | Pre dose to up to 4 hours post dose
Time to Maximum Observed Plasma Concentration (Tmax) of CNTX-3001 | Pre dose to up to 4 hours post dose
Area Under the Concentration-time Curve up to the Last Measurable Concentration of CNTX-3001 | Pre dose to up to 4 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Neurovations, Napa, California, United States